CLINICAL TRIAL: NCT02483884
Title: An Open-label, Multi Center PET/CT Study for Investigation of Safety and Diagnostic Performance of the 68Ga Labeled PET Tracer [68Ga]RM2 in Patients With Primary Prostate Cancer
Brief Title: PET/CT Imaging Study of the Safety and Diagnostic Performance of [68Ga]RM2 in Patients With Primary Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RM2-01-01-14; 2014-003027-21 (EudraCT Number)
Record Dates: First submitted 2015-06-11; First posted 2015-06-29 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: Bombesin; Gastrin-Releasing Peptide; Prostatic Neoplasms; Genital Diseases, Male; Genital Neoplasms, Male; Neoplasms; Neoplasms by Site; Urogenital Neoplasms; Gastrointestinal Agents; Molecular Mechanisms of Pharmacological Action; Neurotransmitter Agents; Pharmacologic Actions; Physiological Effects of Drugs; Therapeutic Uses
MeSH Terms: conditions — Prostatic Neoplasms; Genital Diseases, Male; Genital Neoplasms, Male; Neoplasms; Neoplasms by Site; Urogenital Neoplasms | interventions — BAY 86-7548

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low risk for recurrence (Experimental): Diagnostic [68Ga]RM2 is administered to 10 primary prostate cancer patients with low risk of recurrence who undergo PET/CT 60 min post i.v. for at least 20 min.
  Interventions: Drug: [68Ga]RM2; Procedure: PET/CT
- Intermediate risk for recurrence (Experimental): Diagnostic [68Ga]RM2 is administered to 10 primary prostate cancer patients with intermediate risk of recurrence who undergo PET/CT 60 min post i.v. for at least 20 min.
  Interventions: Drug: [68Ga]RM2; Procedure: PET/CT
- High risk for recurrence (Experimental): Diagnostic [68Ga]RM2 is administered to 10 primary prostate cancer patients with high risk of recurrence who undergo PET/CT 60 min post i.v. for at least 20 min.
  Interventions: Drug: [68Ga]RM2; Procedure: PET/CT

INTERVENTIONS:
Drug: [68Ga]RM2 — [68Ga]RM2 is a novel 68Ga labeled, radiopharmaceutical agent for PET imaging. It is administered intravenously as a single dose of 140 MBq (corresponding to ≤ 40 μg mass dose)
  Other Names: [68Ga] labeled Bombesin derivative; Gallium Ga68-labeled GRPR antagonist RM2
Procedure: PET/CT — Patients received [68Ga]RM2 undergo PET/CT 60 min p.i. for at least 20 min

SUMMARY:
The aim of this study is to investigate safety and diagnostic performance of the 68Ga labeled PET tracer [68Ga]RM2 for detection and localization of primary prostate cancer confirmed by histopathology of the prostate as a standard of truth.

This is an open-label, multi center PET/CT (positron emission tomography/computed tomography) non-randomized study. The study comprises 2 parts with an interim analysis after Part 1. In Part 1 a total of 30 subjects with biopsy-proven primary prostate cancer will be enrolled. Three strata of patients for the first part will be enrolled based on their pretreatment recurrence risk assessment according to the NCCN guidelines: 10 patients with low, 10 patients with intermediate and 10 patients with high pretreatment risk of recurrence.

DETAILED DESCRIPTION:
For inclusion, the prostate cancer needs to be histologically confirmed and MRI and PET/CT with [18F]-choline (18F-choline is not mandatory) should be available for comparison. Diagnostic [68Ga]RM2 will be injected intravenously into the subjects, and PET/CT imaging performed. Images will be assessed visually and quantitatively. Subjects should be scheduled for subsequent prostatectomy within 4 weeks after PET scan.

Prostate cancer will be confirmed by histopathological step-section analysis following prostatectomy and used as Standard of Truth. Based on the results of the initial 30 patients, an expansion cohort of 50 patients for Part 2 will be enrolled to increase the safety and tolerability database and to further characterize the uptake of [68Ga]RM2 in specific subsets.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients with diagnosis of primary prostate cancer in which prostate cancer is histologically confirmed and results of histology are available.
* Patient with planned prostatectomy (within 4 weeks following the [68Ga]RM2 scan).
* Patient had a MRI, and [18F]-choline PET/CT (when available), for primary detection or staging and the images and the results are available (Note: [18F]-choline PET/CT is optional) or the MRI examination is already scheduled at the time of the screening visit for a date before prostatectomy.
* The MRI and [18F]-choline PET/CT referred to in criterion 5 were performed preferably within not more than 5 days prior to the planned imaging with [68Ga]RM2. The maximum interval between MRI and [18F]-choline PET/CT and treatment with [68Ga]RM2 PET/CT is 6 weeks. However, if required, the MRI examination can also be performed after the [68Ga]RM2 PET/CT, but is already scheduled at the time of the screening visit for a date before prostatectomy.
* No chemotherapy, radiotherapy, biopsy or immune/biologic therapy between MRI and [18F]-choline PET/CT (when performed) and [68Ga]RM2 PET/CT performed or scheduled.

NOTE: If MRI is performed after the [68Ga]RM2 PET/CT, no chemotherapy, radiotherapy, biopsy or immune/biologic therapy between [68Ga]RM2 PET/CT and MRI examination is allowed.

* Recovery (excluding alopecia) from previous surgery, radiation, and chemotherapy
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-2 (see Attachments).
* No clinically relevant deviations in renal function as determined by Cockcroft and Gault method using serum creatinine at screening.
* No malfunction equivalent to CTC (Common toxicity criteria) toxicities grade > 2 of the liver (ALT; bilirubin).
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Concurrent severe and/or uncontrolled and/or unstable medical disease other than prostate cancer (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of [68Ga]RM2, unstable and uncontrolled hypertension, chronic renal or hepatic disease, severe pulmonary disease) which could compromise participation in the study.
* Known sensitivity to the study drug or components of the preparation.
* Patient is in custody by order of an authority or a court of law.
* Patient is a relative of the investigator, student of the investigator or otherwise dependent.
* Patient is participating in another clinical study involving administration of an investigational drug at the same time as well as in the preceding 4 weeks before radiotracer administration. Participation in another clinical study involving administration of an investigational drug has ended within the preceding 4 weeks before radiotracer administration.
* Unwillingness or inability to comply with the protocol.
* Patient fulfils criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the patient's safety.
* Hematological or biochemical parameters that are outside the normal range and are considered clinically significant by the investigator, i.e. CTC (Common toxicity criteria) toxicities grade > 2. Minor deviations in lab parameters that are considered by the evaluating physician to be not clinically significant with respect to safety or interpretation of study results are not considered an exclusion criterion.
* History of significant occupational exposure to ionizing radiation or monitoring of occupational radiation exposure (according to recommendations from current guidelines).
* Donation of blood within 12 weeks or plasmapheresis within 2 weeks before the radiotracer Administration.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of [68Ga]RM2 PET to identify lesions in comparison to whole-mount histopathology (number of histologically verified cancer lesions identified) | 60-80 min post injection

SECONDARY OUTCOMES:
Accumulation and tumor detection-rate | 60-80 min post injection
  Evaluation of [68Ga]RM2 accumulation and tumor detection-rate in patients with low, intermediate and high likelihood of recurrence according to pre-treatment risk stratification (NCCN guidelines).
Accumulation of [68Ga]RM2 in BPH | 60-80 min post injection
  Assessment of the accumulation of [68Ga]RM2 in benign prostate hyperplasia (BPH) areas using whole mount sections of the prostate as standard of truth (SOT)
Proportion of lesions detected by [68Ga]RM2 PET in comparison to MRI and [18F]-choline (whenever available) | 60-80 min post injection
  Comparison of [68Ga]RM2 findings to MRI, and [18F]-choline whenever available ([18F]-choline not mandatory)
Quantitative determination (Standardized Uptake Value [SUV]) of [68Ga]RM2 uptake in cancer lesions, stratified according to risk groups | 60-80 min post injection
  Quantitative comparison of [68Ga]RM2 uptake in patients with low, intermediate or high likelihood of recurrence
Evaluation of SUV threshold | 60-80 min post injection
  Exploratory evaluation of a quantitative (SUV) threshold to distinguish low, intermediate and high risk patients based on comparison with post-surgery histopathology

OTHER OUTCOMES:
Number of patients with adverse events | after signing ICF until 5 days post injection
  Evaluation of safety and tolerability of [68Ga]RM2

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Stephens, MD, PhD, Study Director — Piramal Imaging GmbH
Locations (2):
- Krankenhaus der Barmherzigen Schwestern, Linz, Austria
- Turku PET Centre/Department of Oncology and Radiotherapy, Turku, Finland